CLINICAL TRIAL: NCT03897725
Title: Evaluating The Acceptability and Uptake of PrEP for Adolescent Women in The Deep South
Brief Title: Evaluating The Acceptability and Uptake of Pre-Exposure Prophylaxis (PrEP) for Adolescent Women in The Deep South
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Contract terminated
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Tina Y Simpson, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 000523914
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Adolescent Behavior; HIV/AIDS; PrEP
MeSH Terms: conditions — Adolescent Behavior; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telehealth Intervention (Experimental): Study participants will be randomized into either the control or experimental group. Participants in the intervention group will receive routine care which will follow the schedule from previous adolescent PrEP studies where participants are recommended to follow up at 4, 8, and 12 weeks and then every 3 months following initiation of PrEP. This group will also receive SMS texting every 4 weeks between in-person visits (weeks 16, 20, 28,32, 40, 44) reminding them to pick up their medication. The experimental group will also be seen in follow up every month for the first 3 months and then spaced out to visits every 3 months. The SMS texting will occur every 4 weeks between in-person visits, the experimental group will also have 2 tele-health visits (which will be conducted within a participant's home using an app) that will occur every 4 weeks between each of the traditional in-person visits to provide more frequent monitoring and counseling regarding adherence.
  Interventions: Other: Telehealth Coaching
- Routine Care (No Intervention): The control group will follow the schedule from previous adolescent PrEP studies where participants are recommended to follow up at 4, 8, and 12 weeks and then every 3 months following initiation of PrEP.

INTERVENTIONS:
Other: Telehealth Coaching — Telehealth coaching to promote adherence
  Arms: Telehealth Intervention

SUMMARY:
This project is designed to 1) develop a PrEP implementation plan for a general adolescent clinic. Investigators will develop a replicable implementation plan for providing PrEP to adolescents in a primary care setting; and 2) Determine the acceptability and preliminary effectiveness of a telehealth intervention to promote adherence in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Females between 15 to 21 years old
* Established patients at the Adolescent Health Center
* HIV negative

Exclusion Criteria:

* HIV positive patients
* patients weighing less than 35kg
* patients with creatinine clearance <60 ml/min
* patients with documented osteopenia or osteoporosis or history of pathologic fractures
* patients with previous allergic reactions to either emtricitabine or tenofovir
* patients who are on post-exposure prophylaxis for HIV (they can become eligible after completion of therapy)
* patients with hepatic impairment
* For patients who become pregnant, they may be able to continue on PrEP after a discussion with their obstetrics/gynecology (OB/GYN) provider.

Ages: 15 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to PrEP | 1 year
  Retention of adolescent females in PrEP care (attendance at follow-up visits) and adherence to emtricitabine/tenofovir evidenced by dried blood spot sampling

CONTACTS AND LOCATIONS:
Overall Officials: Tina Simpson, MD, Principal Investigator — University of Alabama at Birminghahm
Locations (1):
- William A. Daniel Adolescent Health Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
See below
Supporting Information: Study Protocol, SAP, ICF
Time Frame: To be determined
Access Criteria: To be determined